CLINICAL TRIAL: NCT00828321
Title: Randomized , 2- Way Crossover, Bioequivalence Study of Ramipril 10 mg Capsule and Altace® Administered as 1 x 10 mg Capsule in Healthy Subjects Under Fasting Conditions
Brief Title: Ramipril 10 mg Capsule in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 40179
Record Dates: First submitted 2009-01-12; First posted 2009-01-23 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalency; Healthy Volunteers
MeSH Terms: interventions — Ramipril

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ramipril 10 mg capsule
- 2 (Active Comparator)
  Interventions: Drug: Altace® 10 mg capsule

INTERVENTIONS:
Drug: Ramipril 10 mg capsule — 1 x 10 mg
  Arms: 1
Drug: Altace® 10 mg capsule — 1 x 10 mg
  Arms: 2

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of ramipril 10 mg capsule (test) versus Altace® (reference), administered as 1 x 10 mg capsule under fasting conditions.

DETAILED DESCRIPTION:
Detailed Description

Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

Outcome: Confidence interval fell within 80-125% therefore met the FDA Bioequivalence criteria; no drug related, serious, unexpected adverse events were reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-childbearing potential female, light smoker of non-smoker 18 years of age and older.
* Capable of consent
* Non-childbearing potential female subject is defined as follows:
* Post-menopausal state: absence of menses for 12 months prior to drug administration or hysterectomy with bilateral oophorectomy at least 6 months prior to drug administration, or
* Surgically sterile: hysterectomy, bilateral oophorectomy, or tubule ligation at least 6 months prior to drud administration.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub- Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant, specifically BUN, serum creatinine and hyperkalemia.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* EcG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 100 or over 140 mmHg, diastolic blood pressure lower than 60 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) or change in the systolic blood pressure of 20 mmHg, or diastolic blood pressure of 10mmHg when passing from supine (after at least 5 minutes) to standing position ( after 1-3 minutes), at screening.
* BMI ≥30.0kg/m2.
* History of significant alcohol abuse within 6 months prior to the screening visit of any indication of the regular use of more than 14 units of alcohol per week ( 1 Unit= 150 mL of wine, 360 mL of beer, or 45 mL of 40% hard alcohol), or positive alcohol breath test at screening.
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to the screening visit of hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit of positive urine drug screen at screening.
* History of allergic reactions to heparin, ramipril, or other ACE inhibitors, or other related drugs.
* Use of any drugs known to induce hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoine, glucocorticoids, omeprazole; examples of inhibitors: antidepressant (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of and investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver of kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of hte drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication ( including hormone replacement therapy) within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Smoking more than 10 cigarettes per day.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 30 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* Intolerance to venipunctures
* Clinically significant history of renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will nor be eligible for this study.
* Unable to understand or unwilling to sign the Informed Consent Form.
* Clinically significant history of angioedema.
* History of known presence of volume-depletion (diuretics, dialysis, gastrointestinal disease) or hypotension.
* History of collagen-vascular disease and/or renal disease.
* History of ischemic heart disease, congestive heart failure, or cerebrovascular disease.
* Breast-feeding subject.
* Positive urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — Anapharm
Locations (2):
- Canada (2):
  - Anapharm Inc., Montreal, Quebec
  - Anapharm Inc., Sainte-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Ramipril) First: 10 mg Ramipril Capsules test product dosed in first period followed by 10 mg Altace® Capsules reference product dosed in the second period.
- Reference (Altace®) First: 10 mg Altace® Capsules reference product dosed in first period followed by 10 mg Ramipril Capsules test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Ramipril) First | Reference (Altace®) First
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout of 42 Days
Arm/Group | Test (Ramipril) First | Reference (Altace®) First
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention
Arm/Group | Test (Ramipril) First | Reference (Altace®) First
Started | 18 | 20
Completed | 18 | 19
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Ramipril) First | Reference (Altace®) First | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 0 | 2 | 2
  White | 18 | 17 | 35
  Hispanic | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)of Ramipril
Description: Bioequivalence based on Cmax of Ramipril.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Test (Ramipril): 10 mg Ramipril Capsules test product dosed in either period.
- Reference (Altace®): 10 mg Altace® Capsules reference product dosed in either period.
Arm/Group | Test (Ramipril) | Reference (Altace®)
Number analyzed (Participants) | 37 | 37
pg/mL | 24243.26 (10801.83) | 25646.69 (10793.02)
Statistical Analysis 1: Comparison: Test (Ramipril) vs Reference (Altace®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 94.16, 90% CI [85.08 to 104.21] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)of Ramipril
Description: Bioequivalence based on AUC0-t of Ramipril.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Ramipril) | Reference (Altace®)
Number analyzed (Participants) | 37 | 37
pg*h/mL | 20716.92 (8241.81) | 20859.98 (9796.3)
Statistical Analysis 1: Comparison: Test (Ramipril) vs Reference (Altace®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.22, 90% CI [96.21 to 108.6] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)of Ramipril.
Description: Bioequivalence based on AUC0-t for Ramipril.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Ramipril) | Reference (Altace®)
Number analyzed (Participants) | 37 | 37
pg*h/mL | 21310.07 (8422.26) | 21406.11 (9997.76)
Statistical Analysis 1: Comparison: Test (Ramipril) vs Reference (Altace®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.22, 90% CI [96.34 to 108.58] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)of Ramiprilat.
Description: Informational comparison of Cmax values for the metabolite Ramiprilat.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Test (Ramipril) | Reference (Altace®)
Number analyzed (Participants) | 37 | 37
pg/mL | 25892.38 (17462.37) | 26154.13 (18380.56)
Statistical Analysis 1: Comparison: Test (Ramipril) vs Reference (Altace®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 98.52, 90% CI [92.63 to 104.79] — This analysis was for informational purposes and was not used to establish bioequivalence

5. Secondary Outcome: AUC0-72 (Area Under the Concentration-time Curve From Time Zero to Time 72 Hours)of Ramiprilat.
Description: Informational comparison of AUC0-72 values for the metabolite Ramiprilat.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Ramipril) | Reference (Altace®)
Number analyzed (Participants) | 37 | 37
pg*h/mL | 196669.75 (69676.68) | 201747.51 (73592.98)
Statistical Analysis 1: Comparison: Test (Ramipril) vs Reference (Altace®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.45, 90% CI [94.66 to 100.32] — This analysis was for informational purposes only and was not used to establish bioequivalence

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.